CLINICAL TRIAL: NCT05022407
Title: Impact of COVID-19 Epidemic on Clinical Outcomes and Service Delivery Among People Living With HIV and Health Care Workers in Mozambique
Brief Title: COVID-19 and HIV in Health Workers in Mozambique
Acronym: COVIV
Status: Completed | Type: Observational
Sponsor: Instituto Nacional de Saúde, Mozambique (Other Government)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: CGH-MOZ-9/24/20-ef1f9
Record Dates: First submitted 2021-08-25; First posted 2021-08-26 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Hiv; Covid19
Keywords: HIV; COVID-19; SARS-COV-2
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — If participants have a positive rapid test or are considered eligible for RNA-PCR SARS-CoV-2 testing, 10mL (mililliters) of venous blood (6mL EDTA and 4mL serum tubes) will be collected as stored samples for future research related to COVID-19.
  All participants will have DBS sample collected.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Cohort 1 (SARS-CoV-2 uninfected): Participants who test negative on the SARS-CoV-2 rapid test and are not considered at risk of COVID-19 or who have a negative RNA-PCR SARS-CoV-2 test result at baseline.
- Cohort 2 (SARS-CoV-2 infected): Participants who test positive on RNA-PCR SARS-CoV-2.
- Cohort 3 (SARS-CoV-2 exposed): Participants who have a positive SARS-CoV-2 rapid test result and are not considered to be at risk of active COVID-19 infection or have a negative RNA-PCR SARS-CoV-2 test.
- Cohort 4 ( Vaccinated): Participants who declare having received at least one dose of COVID-19 vaccine (verbally or by showing vaccination card) at inclusion (for HCW or PLHIV) or at any follow-up visit (PLHIV) will be followed in this cohort.

SUMMARY:
While COVID-19 (coronavirus disease 2019) is an important emergent issue for all in the country, there is a significant number of people in the population who are especially vulnerable to the potential impact that the novel coronavirus epidemic may have on their health. The overall purpose of the study is to investigate: (1) the dynamics of COVID-19 infection among people living with HIV and health care workers providing HIV services; (2) the provision of HIV and HIV/TB care and treatment services at health facilities, within the scope of COVID-19 or in the context of COVID-19 and; (3) the perceptions of COVID-19 and access to care among people living with HIV and health care workers providing HIV services.

DETAILED DESCRIPTION:
The protocol is designed to assess prevalence and incidence of COVID-19 among PLHIV and health care workers. Additionally, we aim to evaluate the effect of the COVID-19 epidemic on clinical and immunological outcomes and health care service delivery among PLHIV and HCWs providing HIV services in Mozambique, as well as monitoring breakthrough infections after vaccination. This will facilitate timely estimates of transmissibility of SARS-CoV-2, and of the severity of COVID-19 infection among PLHIV and HCWs providing HIV services, as well as inform public health responses to these vulnerable populations. In Mozambique, this is particularly important as health systems are operating at capacity, and resources to expand services in the country are limited. It is in this context that a novel respiratory pathogen, SARS-CoV-2, could have a potentially severe impact in Mozambique among its estimated 2.2 million HIV-infected persons and the health care providers caring for them. The study protocol will be implemented at national level in up to 11 provinces of Mozambique. Results will be used primarily for program improvement and strengthening and will support the Ministry of Health in the decision making on strategies for the COVID-19 response.

Goal The overarching goal of this protocol is to determine the incidence, prevalence, and clinical manifestations of SARS-CoV-2 among patients living with HIV and healthcare workers providing HIV services, and to assess the knowledge, attitudes and practices (KAP) and the impact that COVID-19 has on them and on the healthcare system.

Objectives Primary Objectives

1. To determine the incidence and prevalence of SARS-CoV-2 among unvaccinated PLHIV enrolled in care.
2. To describe the knowledge, attitudes, practices and perceived risks (KAP-P) regarding SARS-CoV-2, prevention, transmission, and management among PLHIV and HCWs providing HIV services.
3. To evaluate the effect of COVID-19 pandemic on retention to HIV care.

Secondary Objectives

1. To determine the clinical, immunologic, and virological outcomes of SARS-CoV-2 infection in PLHIV and HCWs providing HIV care.
2. To describe the perceptions of PLHIV and HCWs providing HIV services regarding the influence that the COVID-19 pandemic has on the delivery of essential services (including HIV/TB care).
3. To measure the fidelity of participating health facilities to the implementation of national COVID-19 guidelines.
4. To describe COVID-19 breakthrough infection among vaccinated PLHIV and health care workers (HCW) providing HIV care.

ELIGIBILITY:
Inclusion Criteria:

1. PLHIV enrolled in HIV care

   * Have HIV infection and currently in follow-up care at selected HFs;
   * Aged 18 years or older;
   * Able and willing to give informed consent;
   * Willing to test for exposure to SARS-CoV-2 or COVID-19 infection;
   * Willing to be followed and to comply with study visits during the maximum of 15-month study period;
   * Does not intend to move from their residence (requiring change of health facility for HIV care) during the study period;
   * Willing and able to provide contact information.
2. HCWs offering HIV services

   * HCWs (medical doctor, medical officer ["técnico de medicina"], general nurse ["agente de medicina"], maternal and child health [MCH] nurse, pharmacist, laboratory worker, counselor, ancillary worker [e.g., archivist, receptionist], and health volunteers based at the health facility) who are employed full-time and offering HIV services at selected HFs;
   * ≥18 years of age ;
   * Able and willing to give informed consent;
   * Be vaccinated with at least one dose against COVID-19 (verbally or vaccination card));
   * Willing to test for exposure to SARS-CoV-2/ COVID-19 infection;
   * Willing to be followed and available during the maximum of 15-month study period;
   * Does not intend to transfer to another HF during the study period;
   * Willing and able to provide contact information.

Exclusion Criteria:

1. PLHIV enrolled in HIV care

   * Any clinical or mental condition that, in the investigator's opinion, would preclude provision of informed consent or make study participation unsafe or unethical;
   * Any Differentiated Service Delivery where patients have an ART pick-up scheduled less frequently than four times a year (e.g., Community Adherence Support Group [CASG] member);
   * Patients whose antiretroviral (ARV) drugs are picked up by a confidant during their scheduled appointment.
2. HCWs offering HIV services

   * Any clinical or mental conditions that, in the opinion of the investigator or designee, would preclude provision of informed consent or make study participation unsafe or unethical;
   * Individuals working in the HF but from the following cadres: drivers, security personnel, and community health workers/volunteers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1. PLHIV enrolled in HIV care on selected Health facilities.
  2. HCWs offering HIV services in selected Health facilities.
Sampling Method: Probability Sample
Enrollment: 3231 (Actual)
Dates: Start 2021-07-15 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Disease Severity | month 6
  Any disease severity considered as any with severe or critical disease, as per WHO definition.

CONTACTS AND LOCATIONS:
Overall Officials: Edna Viegas, MD, PhD, Principal Investigator — INS-CISPOC
Locations (1):
- INSMozambique, Maputo, Mozambique

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] De Schacht C, Nhacule E, Belo C, Young PW, Bhatt N, Junior F, Pimentel De Gusmao E, Muquingue H, Muteerwa A, Bila D, Ouenzar MA, Madede T, Cumbane R, Amorim G, Viegas E; COVIV Study Collaborative Group. Measuring the burden of SARS-CoV-2 infection among persons living with HIV and healthcare workers and its impact on service delivery in Mozambique: protocol of a prospective cohort study. BMJ Open. 2023 Jun 6;13(6):e068988. doi: 10.1136/bmjopen-2022-068988. PMID 37280029